CLINICAL TRIAL: NCT02092649
Title: Effects of 12 Weeks of Omega 3 Supplementation on Resting Metabolic Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Lawrence Spriet, Professor and Chair, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14JA044
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Whole Body Energy Metabolism
Keywords: Omega-3; Resting metabolic rate; Eicosapentaenoic acid; Docosahexaenoic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Complete (Experimental): Oral ingestion of 3000 mg (5 capsules) of Omega-3 Complete (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks.
  Interventions: Dietary Supplement: Omega-3 Complete
- Placebo Pill (Placebo Comparator): Oral ingestion of 3 capsules of a placebo olive oil pill (Swanson Health Products, PO Box 2803 - Fargo, ND 58108 USA) per day for 12 weeks.
  Interventions: Dietary Supplement: Placebo Pill

INTERVENTIONS:
Dietary Supplement: Omega-3 Complete
  Arms: Omega-3 Complete
Dietary Supplement: Placebo Pill
  Arms: Placebo Pill

SUMMARY:
Fatty acids are the main components of the cell membranes. It has been demonstrated that diet can alter the characteristics and function of many membranes in the body, which has an effect on cardiovascular and metabolic health. Over the last two decades there has been a substantial rise in the research of the effects of Omega 3 polyunsaturated fatty acids on bodily function. There are two fatty acids that are of particular interest to researchers, eicosapentanoic acid (EPA) and docosahexanoic acid (DHA). These fatty acids have unique unsaturated structures, and their incorporation into biological membranes seems to generate important and positive physiological effects. The body is unable to synthesize these fatty acids in high concentrations to elicit significant effects, so they must be obtained through diet in food or via supplementation.

It has been suggested that EPA and DHA supplementation increases resting metabolic rate (RMR) in humans, in part by increasing the use of fat as a fuel during rest. There are a limited number of studies examining the effects of Omega 3 supplementation on RMR. Some have found an increase in RMR while others have found no change. These studies have some limitations, as that they have either used a small sample size, a low omega fatty acid dose and/or short supplementation periods. Due to the variable results, the investigators will improve the reliability of the RMR measurements by making measures on each subject during two consecutive days at each time point that it is measured (0, 6 and 12 weeks).

Therefore, the purpose of this study is to determine the effects of 12 weeks of omega 3 supplementation (3 g/d) on healthy young adults vs. the supplementation of a placebo. The researchers hypothesize that EPA and DHA supplementation will result in an increase in RMR and fat oxidation in some subjects and not in others. The duplicate RMR measures will determine the prevalence and magnitude of the omega 3 supplementation.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years of age.
* Must currently practice a consistent diet and exercise regimen, and maintain this throughout the duration of the study.

Exclusion Criteria:

* Current or previous supplementation with omega-3's.
* Average fish intake greater than two times per week.
* Taken any medications, have any medical condition, and hospitalization or surgeries.
* Allergy to fish/fish oil, , (rosemary extract, ascorbyl palmitate, or natural tocopherols).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence L Spriet, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Jannas-Vela S, Roke K, Boville S, Mutch DM, Spriet LL. Lack of effects of fish oil supplementation for 12 weeks on resting metabolic rate and substrate oxidation in healthy young men: A randomized controlled trial. PLoS One. 2017 Feb 17;12(2):e0172576. doi: 10.1371/journal.pone.0172576. eCollection 2017. PMID 28212390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: May 2014 - Dec 2014 Location: University of Guelph
Groups:
- Omega-3 Complete: Oral ingestion of 3000 mg (5 capsules) of Omega-3 Complete (Jamieson Laboratories Ltd., Windsor, Ontario, Canada) per day for 12 weeks.
  Omega-3 Complete
- Placebo Pill: Oral ingestion of 3 capsules of a placebo olive oil pill (Swanson Health Products, PO Box 2803 - Fargo, ND 58108 USA) per day for 12 weeks.
  Placebo Pill
Period: Overall Study
Arm/Group | Omega-3 Complete | Placebo Pill
Started | 13 (13 participants recruited) | 13 (13 participants recruited)
Completed | 13 (13 participants finished study) | 13 (13 participants finished study)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We expect to have a normal distribution of participants in both groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Complete | Placebo Pill | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (3.29) | 22 (1.61) | 23 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 13 | 26
Resting Metabolic Rate [Mean (Standard Deviation); unit: kcal/day] | 2041 (187) | 2016 (227) | 2029 (204)

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Metabolic Rate From Baseline
Description: Percent change in resting metabolic rate
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 13 | 13
percent change
  Baseline - Week 6 | -0.19 (4.70) | -0.19 (4.70)
  Baseline - Week 12 | 0.67 (8.65) | 1.11 (6.51)

2. Secondary Outcome: Change in Maximum Oxygen Consumption From Baseline
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 13 | 13
percent change | 3.30 (5.54) | 2.17 (5.52)

3. Secondary Outcome: Change in Whole Body Resting Fat Oxidation From Baseline
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 13 | 13
percent change
  Baseline - Week 6 | 0.39 (34.53) | 2.92 (31.37)
  Baseline - Week 12 | 19.52 (38.39) | 17.82 (48.56)

4. Secondary Outcome: Change in Whole Body Resting Carbohydrate Oxidation From Baseline
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 13 | 13
percent change
  Baseline - Week 6 | -3.47 (42.05) | 7.23 (32.64)
  Baseline - Week 12 | -12.41 (39.15) | 14.23 (42.86)

5. Secondary Outcome: Variability of Resting Metabolic Rate Measurement on 2 Consecutive Days
Time Frame: Baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percent variability
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 13 | 13
percent variability
  Week 0 | 2.70 (2.44) | 2.57 (1.32)
  Week 6 | 3.98 (3.30) | 2.77 (2.04)
  Week 12 | 3.22 (2.97) | 2.18 (1.82)

6. Secondary Outcome: Change in Fasted Blood Triglyceride Concentration From Baseline
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omega-3 Complete | Placebo Pill
Number analyzed (Participants) | 12 | 12
percent change | -18.07 (44.44) | -2.41 (60.00)

ADVERSE EVENTS:
Arm/Group | Omega-3 Complete | Placebo Pill
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No